CLINICAL TRIAL: NCT00798967
Title: A 24-Week Study of the Efficacy and Safety of Teduglutide in Subjects With Parenteral Nutrition-Dependent Short Bowel Syndrome
Brief Title: Study of Teduglutide Effectiveness in Parenteral Nutrition (PN)-Dependent Short Bowel Syndrome (SBS) Subjects
Acronym: STEPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Nycomed (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL0600-020; 2008-006193-15 (EudraCT Number)
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Short Bowel Syndrome
Keywords: SBS; short bowel syndrome; TPN; parenteral nutrition; PN
MeSH Terms: conditions — Short Bowel Syndrome; Hyperphagia | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teduglutide (Experimental): 0.05 mg/kg/day sc dose of teduglutide
  Interventions: Drug: teduglutide
- Placebo (Placebo Comparator): Matching subcutaneous dose of placebo to teduglutide
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: teduglutide — 0.05 mg/kg/day sc injection for 24 weeks
  Other Names: GATTEX; ALX-0600
  Arms: Teduglutide
Drug: placebo — Matching daily subcutaneous dose of placebo to teduglutide for 24 weeks
  Arms: Placebo

SUMMARY:
Teduglutide is an investigative medicine being evaluated as a possible treatment for people with parenteral nutrition (PN) dependent Short Bowel Syndrome (SBS). Teduglutide is similar to a protein the body makes. When people have SBS, their bodies do not make enough of the protein and they have trouble getting nutrients and fluids from the food they eat and drink. This study was designed to provide evidence of efficacy, safety, and tolerability of teduglutide 0.05 mg/kg daily in SBS subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to any study-related procedures are performed
* Men and women 18 years of age or older at the time of informed consent signing
* Intestinal failure resulting in Short Bowel Syndrome
* At least 12 months of continuous PN dependency
* 12 weeks of clinical remission of Crohn's disease (CD) prior to dosing
* PN required at least 3 times weekly
* A stable PN volume for four weeks prior to dosing

Exclusion Criteria:

* History of cancer or clinically significant lymphoproliferative disease with fewer than 5 years documented disease-free state
* Participation in clinical study within 30 days for drug or 90 days for antibody
* Use of native GLP-2 or human growth hormone (HGH) within 6 months of screening
* Use of iv glutamine within 30 days prior to screening
* Use of teduglutide
* CD patients who have been treated with biological therapy within 6 months of screening
* IBD patients who require chronic systemic immunosuppressant therapy
* More than 4 SBS- or PN-related hospitalizations within 12 months of screening
* Unplanned hospitalization within one month of screening
* Pregnant or lactating women
* Body weight > 88kg
* Body mass index (BMI) < 15 kg/m2
* Severe hepatic impairment or disturbed renal function
* Female subjects who are not surgically sterile or postmenopausal or who are not using medically acceptable methods of birth control during and for 30 days after the treatment period
* Not capable of understanding or not willing to adhere to the study visit schedules and other protocol requirements
* Any condition or circumstance that is the investigator's opinion would put the subject at any undue risk, prevent completion of the study, or interfere with the analysis of the study results
* Significant active, uncontrolled, untreated systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-11-25 (Actual); Primary Completion 2011-01-25 (Actual); Study Completion 2011-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (35):
- United States (11):
  - Scripps Clinic & Research Foundation, La Jolla, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - Mount Sinai Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennslyvania, Philadelphia, Pennsylvania
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (4):
  - Critical Care Research, Royal Alexandra Hospital, Edmonton, Alberta
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Polyclinic Family and Specialty Medicine Facility, North York, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
- Rigshospitalet - Abdominalcentret, Hepatologisk Kilinik A, Copenhagen, Denmark
- France (3):
  - Hôpital Beaujon, Clichy
  - Hôpital Croix Rousse Unité de Nutrition Clinique Intensive, Lyon
  - Hôpital de l'Archet Pôle Digestif, Nice
- Germany (3):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Israelitisches Krankenhaus, Hamburg, Hamburg
  - Med. Klinik m.S. Hepatologie und Gastroenterologie, Berlin, State of Berlin
- Italy (3):
  - Azienda Ospedaliera Universitaria S. Giovanni Battista - Le Molinette, Torino, TO
  - Policlinico Sant'Orsola - Malpighi centro insufficienza intestinale, Bologna
  - Azienda Universitaria Policlinico Federico II, Napoli
- Universitair Medisch Centrum St. Radboud, Nijmegen, Netherlands
- Poland (4):
  - Wojewodzki Szpital Specjalistyczny im. M. Pirogowa, Pracownia Leczenia Zywieniowego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Klinika Chirurgii Ogolnej i Transplantacyjnej, Lublin
  - Wojewodzki Szpital Specjalistyczny,, Olsztyn
  - Samodzielny Publiczny Szpital Kliniczny im. prof W. Orlowskiego CMKP, Oddzial Kliniczny Zywienia i Chirurgii, Warsaw
- Spain (2):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (3):
  - St. Mark's Hospital Northwick Park, Harrow, GT LON
  - University College Hospital, London, GT LON
  - Green Area, Main Hospital Salford Royal Hospitals NHS Foundation Trust, Manchester, GT MAN

REFERENCES:
- [Result] Jeppesen PB, Sanguinetti EL, Buchman A, Howard L, Scolapio JS, Ziegler TR, Gregory J, Tappenden KA, Holst J, Mortensen PB. Teduglutide (ALX-0600), a dipeptidyl peptidase IV resistant glucagon-like peptide 2 analogue, improves intestinal function in short bowel syndrome patients. Gut. 2005 Sep;54(9):1224-31. doi: 10.1136/gut.2004.061440. PMID 16099790
- [Derived] Jeppesen PB, Gabe SM, Seidner DL, Lee HM, Olivier C. Citrulline correlations in short bowel syndrome-intestinal failure by patient stratification: Analysis of 24 weeks of teduglutide treatment from a randomized controlled study. Clin Nutr. 2020 Aug;39(8):2479-2486. doi: 10.1016/j.clnu.2019.11.001. Epub 2019 Nov 9. PMID 31784300
- [Derived] Jeppesen PB, Gabe SM, Seidner DL, Lee HM, Olivier C. Factors Associated With Response to Teduglutide in Patients With Short-Bowel Syndrome and Intestinal Failure. Gastroenterology. 2018 Mar;154(4):874-885. doi: 10.1053/j.gastro.2017.11.023. Epub 2017 Nov 22. PMID 29174926
- [Derived] Fujioka K, Jeejeebhoy K, Pape UF, Li B, Youssef NN, Schneider SM. Patients With Short Bowel on Narcotics During 2 Randomized Trials Have Abdominal Complaints Independent of Teduglutide. JPEN J Parenter Enteral Nutr. 2017 Nov;41(8):1419-1422. doi: 10.1177/0148607116663481. Epub 2016 Aug 9. PMID 27507402
- [Derived] Vipperla K, O'Keefe SJ. Study of teduglutide effectiveness in parenteral nutrition-dependent short-bowel syndrome subjects. Expert Rev Gastroenterol Hepatol. 2013 Nov;7(8):683-7. doi: 10.1586/17474124.2013.842894. Epub 2013 Oct 17. PMID 24134154
- [Derived] Jeppesen PB, Pertkiewicz M, Forbes A, Pironi L, Gabe SM, Joly F, Messing B, Loth S, Youssef NN, Heinze H, Berghofer P. Quality of life in patients with short bowel syndrome treated with the new glucagon-like peptide-2 analogue teduglutide--analyses from a randomised, placebo-controlled study. Clin Nutr. 2013 Oct;32(5):713-21. doi: 10.1016/j.clnu.2013.03.016. Epub 2013 Mar 28. PMID 23587733
- [Derived] Berghofer P, Fragkos KC, Baxter JP, Forbes A, Joly F, Heinze H, Loth S, Pertkiewicz M, Messing B, Jeppesen PB. Development and validation of the disease-specific Short Bowel Syndrome-Quality of Life (SBS-QoL) scale. Clin Nutr. 2013 Oct;32(5):789-96. doi: 10.1016/j.clnu.2012.12.001. Epub 2012 Dec 12. PMID 23274148
- [Derived] Jeppesen PB, Pertkiewicz M, Messing B, Iyer K, Seidner DL, O'keefe SJ, Forbes A, Heinze H, Joelsson B. Teduglutide reduces need for parenteral support among patients with short bowel syndrome with intestinal failure. Gastroenterology. 2012 Dec;143(6):1473-1481.e3. doi: 10.1053/j.gastro.2012.09.007. Epub 2012 Sep 11. PMID 22982184
- See also: HPN support — http://www.oley.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Screened - November 25, 2008; Last Patient Screened - July 13, 2010; First Patient Randomized - March 3, 2009; Last Patient Randomized - July 22, 2010; Locations - hospitals and transplant centers; Subjects must be on parenteral nutrition (PN) and/or intravenous (I.V.) fluids.
Pre-assignment Details: Stage 1 was screening, optimization, and stabilization periods. At screening, if the PN/I.V. volume is not stable per protocol, s/he entered an optimization period (up to 8 weeks) to find the minimally tolerated stable volume of PN/I.V.. Prior to randomization, all entered 4-8 weeks of stabilization period on that volume of PN/I.V.
Groups:
- Teduglutide: 0.05 mg/kg/day subcutaneous (sc) dose of teduglutide
- Placebo: Matching sc dose of placebo to teduglutide
Period: Overall Study
Arm/Group | Teduglutide | Placebo
Started | 43 | 43
Discontinued During Dosing Period | 4 | 4
Completed | 39 | 39
Not Completed | 4 | 4
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Randomized in error by site | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teduglutide | Placebo | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.6) | 49.7 (15.6) | 50.3 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Responder
Description: Comparison of subjects treated with teduglutide to placebo who achieve a 20 to 100% reduction from baseline in weekly parenteral nutrition/intravenous fluid (PN/I.V.) volume at weeks 20 and 24.
Time Frame: Weeks 20 and 24
Population: Percentages were based on the number of subjects in the Intent to Treat (ITT) population.
Measure: Number; unit: subjects
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 43 | 43
subjects | 27 | 13
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) test adjusted for the randomization stratification variable (<= 6 or > 6 L/week of PN at baseline)

2. Secondary Outcome: Absolute Change in PN/I.V. Volume From Baseline to Last Time Point
Description: Absolute change in the volume of PN/I.V. from baseline (Week 0) to the visit when the last data point was collected (week 4 through week 24, or earlier if the subject discontinued early).
Time Frame: Week 0 to last visit when data was collected.
Population: Intent-to-Treat (ITT) was defined for efficacy analyses which included all randomized patients.
Measure: Mean (Standard Deviation); unit: Liters/Week
Arm/Group | Teduglutide | Placebo
Number analyzed (Participants) | 40 | 43
Liters/Week | -4.28 (3.81) | -2.38 (2.79)
Statistical Analysis 1: Comparison: Teduglutide vs Placebo; Last Dosing Visit; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each subject from the time informed consent was signed to end of study. For this reporting of adverse event, the most commonly reported treatment emergent adverse events (>=3 subjects at SOC level) are listed.
Description: All adverse experience reporting used the Safety population which consisted of 85 subjects who received at least one dose of study drug. There were 42 subjects treated with teduglutide, whereas 43 subjects received placebo. Adverse experience monitoring was performed through investigator assessment and safety laboratory testing at every visit.
Arm/Group | Teduglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 15/42 | 12/43
Other Adverse Events (participants affected / at risk) | 35/42 | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (N=42) | Placebo (N=43)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 3 (3)
Catheter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Catheter-related complication (General disorders) | 1 (1) | 0 (0)
Catheter-related infection (Infections and infestations) | 5 (5) | 1 (1)
Central line infection (Infections and infestations) | 2 (2) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Device breakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Implant site extravasation (General disorders) | 1 (1) | 1 (1)
Infective thrombosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (N=42) | Placebo (N=43)
Abdominal distension (Gastrointestinal disorders) | 9 (14) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (14) | 10 (14)
Central line systemic infections (Infections and infestations) | 7 (12) | 7 (8)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 5 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Edema peripheral (General disorders) | 7 (8) | 2 (3)
Fatigue (General disorders) | 4 (5) | 3 (3)
Flatulence (Gastrointestinal disorders) | 5 (5) | 3 (3)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 10 (11) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (19) | 8 (12)
Pyrexia (General disorders) | 4 (5) | 4 (5)
Urinary tract infection (Infections and infestations) | 6 (6) | 4 (5)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (10)
Weight increased (Investigations) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of NPS Pharmaceuticals agreements with its investigators may vary. However, NPS does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.